CLINICAL TRIAL: NCT00977041
Title: Neurofeedback Treatment of Pain in Persons With SCI: Phase 2
Brief Title: Neurofeedback Treatment of Pain in Persons With Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Mark Jensen, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36292-D Phase 2; 124155
Record Dates: First submitted 2009-07-27; First posted 2009-09-15 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Cord Injuries; Pain
Keywords: Neurofeedback
MeSH Terms: conditions — Spinal Cord Injuries; Pain | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurofeedback (Experimental): See Intervention description below.
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — Electrodes will be placed over the temporal lobes bilaterally and a ground electrode placed on the left earlobe. EEG activity will be amplified using a Procomp 2 or Nexus amplifier, and EEGer software will be used to provide subjects with feedback. Contingencies will be set such that alpha brain activity will be reinforced, and high beta and theta brain activity will be inhibited. Standard NF training procedures will be used, which involve simply asking subjects to relax while looking at the feedback screen and "Do whatever is necessary to make and keep the bar wide." This protocol will be repeated for up to 40 60-minute sessions (that will include 30 minutes of NF training), scheduled at least weekly.

SUMMARY:
A number of studies suggest that training to increase different types of brain waves is related to pain relief. The purpose of the second phase of this study is to see if neurofeedback training might help people with chronic pain control their pain better. The information from the study may help the investigators treat chronic pain better in the future.

DETAILED DESCRIPTION:
During this phase of the study, research personnel will provide up to 15 of the subjects with SCI-related pain with a full course (up to 40 sessions) of NF training to determine the effects of this treatment on (a) chronic daily pain, (b) EEG-assessed frequency band amplitudes, and (c) other measures of quality of life (specifically, sleep quality, fatigue, and pain interference).

Standard NF training procedures will be used that involve simply asking participants to relax while looking at the feedback screen and to "Do whatever is necessary to make and keep the color bar wide." EEG bandwidth activity that is associated with being pain-free or with experiencing less pain will be reinforced. This protocol will be repeated for up to 40 30-minute sessions, scheduled at least weekly (but more often if the participant and study PI can arrange this with their schedules. Brain wave activity will be measured three times during the study: once before treatment begins, once immediately after treatment ends, and three months following treatment. Research staff will collect data regarding pain intensity and quality of life from subjects via the telephone three times: before treatment, immediately after treatment, and three months after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older.
2. At least 12 months post-SCI.
3. Otherwise healthy (i.e., no other secondary medical complications, such as pressure ulcers, that could impact pain scores).
4. Read, write and understand English.
5. Experience SCI-related pain on a daily basis.
6. Report an average pain intensity of at least 4 on a 0-10 Numerical Scale.
7. An individual must have one significant pain problem that is the worst or most painful if he/she has more than one pain problem.
8. Pain problem has lasted at least six months, and began after injury.

Exclusion Criteria:

1. History of seizure activity or has non-normative brain activity.
2. Suicidal or paranoid thoughts.
3. Presence of traumatic brain injury or significant skull defects.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Average daily (past 24 hours) pain will be the primary outcome measure for the clinical phase of this study. This will be assessed using a 0-10 NRS via four phone interviews performed on different days by a research assistant. | Just before treatment begins, just after treatment ends (approximately 1 to 6 months following the beginning of treatment), and 3 months following the end of treatment.

SECONDARY OUTCOMES:
Brain wave activity will be assessed in all of second phase participants with the use of an electroencephalogram(EEG). | EEG activity will be collected just before the first treatment session (baseline), just after the last treatment session, and three months following the end of treatment.
Sleep quality will be assessed using the six-item Medical Outcomes Study Sleep measure(Hays & Stewart, 1992). | Just before treatment begins, just after treatment ends (approximately 1 to 6 months following the beginning of treatment), and 3 months following the end of treatment.
Pain interference will be assessed using the PROMIS Pain Impact Scale. | Just before treatment begins, just after treatment ends (approximately 1 to 6 months following the beginning of treatment), and 3 months following the end of treatment.
Fatigue severity will be assessed using the Fatigue Severity Scale (FSS; Krupp et al., 1998). The FSS is a 9-item measure assessing both fatigue severity and impact. | Just before treatment begins, just after treatment ends (approximately 1 to 6 months following the beginning of treatment), and 3 months following the end of treatment.
Medication use in the week prior to each assessment including medication use as well as pain treatments such as massage. | Just before treatment begins, just after treatment ends (approximately 1 to 6 months following the beginning of treatment), and 3 months following the end of treatment.
Benefits received from treatment. | Following the end of treatment (approximately 1 to 6 months after treatment begins) and 3 months following the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Jensen, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Jensen MP, Gertz KJ, Kupper AE, Braden AL, Howe JD, Hakimian S, Sherlin LH. Steps toward developing an EEG biofeedback treatment for chronic pain. Appl Psychophysiol Biofeedback. 2013 Jun;38(2):101-8. doi: 10.1007/s10484-013-9214-9. PMID 23532434